CLINICAL TRIAL: NCT01116336
Title: Phase I Study of Chemoprevention With Green Tea Polyphenon E (PPE) and the Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor Erlotinib (OSI-774, Tarceva) in Patients With Premalignant Lesions of the Head and Neck
Brief Title: Phase I Chemoprevention Trial With Green Tea Polyphenon E & Erlotinib in Patients With Premalignant Lesions of the Head & Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Astellas Pharma Inc (Industry); Polyphenon Pharma (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dong Shin, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00014010; WCI1549-08 (Other: Winship Cancer Institute); 5P50CA128613 (NIH)
Record Dates: First submitted 2010-04-09; First posted 2010-05-05 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Cancer of Head and Neck; Neoplasms, Head and Neck
Keywords: Pre-cancerous conditions; Head and neck tumors; Cancer of head and neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib and Green Tea Polyphenon E (Experimental): Patients will receive erlotinib, at pre-defined dose level, with polyphenon E.
  Interventions: Drug: Erlotinib; Dietary Supplement: Green Tea Polyphenon E

INTERVENTIONS:
Drug: Erlotinib — Participants will be given erlotinib orally (dose escalation from 50 mg, 75 mg, or 100 mg daily continuously for 6 cycles (each cycle is 28 days).
  Other Names: OSI-774; Tarceva
Dietary Supplement: Green Tea Polyphenon E — Participants will also be given PPE orally (200 mg EGCG) three times daily for 6 cycles (each cycle is 28 days). PPE capsules will be taken on a full stomach, within one hour after eating a substantial meal.
  Other Names: EGCG

SUMMARY:
The purpose of this study is to test the preventive effects of a combination of drugs: polyphenon E (PPE) derived from green tea extracts, and erlotinib. Because this combination of drugs has not been tested in humans before for the prevention of cancer, it is not clear which dose of each agent will be optimal in combination.

We will test the safety of the combination of PPE and erlotinib and see what effects (good and/or bad) it has on the patient's premalignant lesion, and find the highest dose of each agent that can be given in combination without causing severe side effects.

ELIGIBILITY:
Inclusion Criteria

* Participants with premalignant lesions (mild dysplasia, moderate dysplasia, severe dysplasia, or carcinoma in situ) of the head and neck, as confirmed by biopsy within the 4 months prior to study entry or a treated primary T1N0 or T2N0 squamous cell carcinoma will be eligible.
* For patients with T1N0 or T2N0 treated squamous cell carcinoma, they must have been free of disease for a minimum period of 8 weeks, up to a maximum of 3 years following completion of surgery and/or radiotherapy.
* Eligible tumor and premalignant lesion sites include oral cavity (buccal mucosal, gingival, floor of mouth, dorsal/ventral tongue, pharyngeal wall), oropharynx, larynx (glottis, supraglottis, subglottis, epiglottis), hypopharynx paranasal sinus and nasal cavity.
* Patients with a treated tumor 1-node 0 (T1N0) or tumor 2-node 0 (T2N0) squamous cell carcinoma may have oral premalignant lesions (i.e., hyperplasia, dysplasia, carcinoma in situ) at the time of study entry (provided their Stage I or II disease has been definitively treated).
* Lesion sites include oral cavity (buccal mucosa, gingival, floor of mouth, dorsal/ventral tongue, pharyngeal wall), oropharynx, hypopharynx,larynx (glottis, supraglottis, subglottis, epiglottis), nasopharynx and paranasal sinuses.
* Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status of 0-1.
* No medical contraindications for flexible laryngoscopy using topical anesthesia, and in the setting of a contraindication to topical anesthesia, general anesthesia may not be used as a substitute.
* General anesthesia, if indicated, is acceptable in patients whose lesions would require general anesthesia for laryngoscopy and biopsy according to routine standard of care.
* Blood counts: total neutrophil count > 1,500/mm³; platelet count > 100,000/mm³.
* Adequate liver function:

  * Total bilirubin level ≤ 1.5 times upper limit normal (ULN)
  * Albumin > 2.5 g/dl
  * Alkaline phosphatase, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN
* Adequate renal function: serum creatinine < 1.5 mg/dl.
* Hemoglobin level ≥ 11gm/dl (age adjusted if appropriate) provided by the reference laboratory performing the test.
* Patients not taking warfarin must have prothrombin time (PT)/partial thromboplastin time (PTT) levels ≤ 1.5 times the upper limit of normal provided by the reference laboratory performing the test.
* Adequate pulmonary function: forced expiratory volume at one second (FEV1) and forced vital capacity (FVC) at least 60% predicted value by spirometry.
* Signed written informed consent.
* The effects of polyphenon E on the developing human fetus at the recommended dose are unknown. For this reason and because polyphenon E may be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.
* Women of child-bearing potential must also have a negative urine pregnancy test (β-HCG) within 72 hours of receiving treatment.
* Must be able to swallow the oral doses of erlotinib and PPE.
* Must be willing to abstain from drinking green tea or taking supplements containing green tea or green tea compounds, for the duration of the investigation and for 30 days prior to study entry.
* Please note that patients with a treated T1N0 or T2N0 squamous carcinoma and who do not have a pre-malignant measurable lesion at the time of study entry will not be subjected to a biopsy but will have cytobrush samples taken as specified in the protocol.

Exclusion Criteria

* Because no dosing or adverse event data are currently available on the use of Polyphenon E in participants < 18 years of age, children are excluded from this study.
* Participants with hyperplasia, in absence of dysplasia or carcinoma in situ, will be excluded because there is possibly no benefit.
* Participants with acute intercurrent illness or those who had surgery within the preceding 4 weeks unless they have fully recovered.
* History of previous malignancies unless the cancer was stage I or II and rendered free of disease more than 1 year.
* Participants who are pregnant or breast feeding. Pregnant women are excluded from this study because Polyphenon E is an investigational agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Polyphenon E, breastfeeding should be discontinued if the mother is treated with Polyphenon E.
* Not practicing adequate contraception if the participants are of child bearing potential.
* Uncontrolled intercurrent illness including, but not limited to, severe active infection, symptomatic congestive heart failure, myocardial infarction within the past six months, unstable angina pectoris, serious cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements are excluded.
* Documented history of coagulopathy such as hemophilia or Von Willebrand's disease or inherited thrombophilia.
* Hypertension not adequately controlled by medication (i.e. systolic blood pressure ≥ 150 and/or diastolic blood pressure ≥ 90 on at least two separate readings).
* History of congestive heart failure (CHF) greater than New York Heart Association (NYHA) Grade II.
* Participants who exhibit confusion, disorientation, or have a history of major psychiatric illness which may impair their understanding of the informed consent.
* Taking epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors within 3 months of study entry.
* Documented history of interstitial lung disease or pulmonary fibrosis.
* Known connective tissue disease.
* Patients who have participated in a clinical trial of an investigational drug within 12 months prior to enrollment.
* History of liver disease or AST and ALT ≥ 2.5 times ULN on screening.
* Consumption of green tea or supplements containing green tea or tea extract within 30 days prior to enrollment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to polyphenon E, tea, or any of the inactive ingredients present in the active or placebo drug products, including gelatin capsules.
* Any condition which would make the subject, in the opinion of the investigator, unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-03; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of erlotinib when administered with a constant dose of green tea polyphenon E (PPE). | Cytobrush/biopsy at three months
  Define MTD as the dose level of erlotinib when administered with a constant dose of 200 mg (EGCG) TID of Green Tea Polyphenon E (PPE) to a patient results in a probability equal to θ = 0.33 that a dose-limiting toxicity (DLT) will be manifest within 1 cycle defined as 28 days.

SECONDARY OUTCOMES:
To assess the safety of the combination of PPE and erlotinib in patients receiving 3 different doses of erlotinib (50 mg, 75 mg, and 100 mg) in combination with PPE (200 mg EGCG TID) for 6 months. | Baseline, 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dong M. Shin, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland